CLINICAL TRIAL: NCT04540744
Title: A Single-center, Open-label, Single-dose, Randomized, 2-way Crossover Phase 1 Study in Healthy Adult Participants to Assess the Relative Oral Bioavailability of the Combination of Macitentan/Tadalafil (10 mg/20 mg) Administered a Fixed-dose Combination Formulation Compared to the Reference Free Combination of 10 mg Macitentan (Opsumit®) and 20 mg Tadalafil (Adcirca®)
Brief Title: A Study of Macitentan/Tadalafil Combination Administered a Fixed-dose Combination Formulation Compared to the Reference Free Combination of Macitentan and Tadalafil
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR108794; 2020-000566-42 (EudraCT Number); 67896062PAH1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-09-02; First posted 2020-09-07 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Healthy
MeSH Terms: interventions — Tadalafil; macitentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Sequence AB (Experimental): Participants will receive a single oral dose of fixed dose combination (FDC) of macitentan/tadalafil (10 milligram [mg]/20 mg) in fasted conditions (test) (Treatment A) in treatment period 1 followed by a single oral dose of a free combination of 10 mg macitentan and 20 mg tadalafil in fasted conditions (reference) (Treatment B) in treatment period 2 on Day 1. Study drug intake in subsequent treatment periods in an individual participant will be separated by a washout period of at least 10 days.
  Interventions: Drug: FDC of macitentan/tadalafil (10 mg/20 mg); Drug: Macitentan 10 mg; Drug: Tadalafil 20 mg
- Treatment Sequence BA (Experimental): Participants will receive Treatment B in treatment period 1 followed by Treatment A in treatment period 2 on Day 1. Study drug intake in subsequent treatment periods in an individual participant will be separated by a washout period of at least 10 days.
  Interventions: Drug: FDC of macitentan/tadalafil (10 mg/20 mg); Drug: Macitentan 10 mg; Drug: Tadalafil 20 mg

INTERVENTIONS:
Drug: FDC of macitentan/tadalafil (10 mg/20 mg) — FDC of macitentan/tadalafil (10 mg/20 mg) tablet will be administered orally as per assigned treatment sequence.
  Other Names: Opsumit; Adcirca
Drug: Macitentan 10 mg — Macitentan 10 mg tablet will be administered orally as a free combination as per assigned treatment sequence.
  Other Names: Opsumit
Drug: Tadalafil 20 mg — Tadalafil 20 mg tablet will be administered orally as a free combination as per assigned treatment sequence.
  Other Names: Adcirca

SUMMARY:
The purpose of this study is to assess the rate and extent of absorption of macitentan and tadalafil following administration of a single oral dose of a fixed-dose combination (FDC) of 10 milligram (mg)/20 mg macitentan/tadalafil (test), compared to the coadministration as a free combination (reference) of 10 mg macitentan and 20 mg tadalafil under fasted conditions in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Must sign an informed consent form (ICF) indicating they understand the purpose of, and procedures required for, the study and are willing to participate in the study, before starting any screening activities
* Body mass index (BMI; weight [kg]/height^2 [m]^2) between 18.5 and 30.0 kilogram per meter square (kg/m^2) inclusive, and body weight not less than 50.0 kg at screening
* Healthy on the basis of physical examination, medical and surgical history, performed at screening. If there are abnormalities, the participant may be included only if the investigator judges the abnormalities to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the investigator
* Systolic blood pressure (SBP) between 100 and 145 millimeter of Mercury (mmHg) (inclusive) and diastolic blood pressure (DBP) between 50 and 90 mmHg (inclusive) at screening, preferably measured on the right arm, supine after 5 minutes of rest and standing after 3 minutes
* Twelve-lead electrocardiogram (ECG) with heart rate between 45 and 90 beats per minute (bpm) and without clinically relevant abnormalities, at the discretion of the investigator, measured after the participant is supine for at least 5 minutes, at screening
* During the study (from the day of first study drug intake onwards) and for a minimum of 1 spermatogenesis cycle (defined as approximately 90 days) after the last study drug intake, a male participant must agree: (a) to wear a condom when engaging in any activity that allows for passage of ejaculate to another person (male participant should also be advised of the benefit for a female partner to use a highly effective method of contraception as condom may break or leak); (b) not to donate sperm for the purpose of reproduction.

Contraceptive use by men or women should be consistent with local regulations regarding the use of contraceptive methods for participants participating in clinical studies

Exclusion Criteria:

* Female participant who is breastfeeding at screening and/or plans to breastfeed throughout the study until 30 days after last study drug intake
* Known allergies, hypersensitivity, or intolerance to any active substance or drugs of the same class, or any excipient of the drug formulation(s)
* Values of hepatic aminotransferase (alanine aminotransferase and/or aspartate aminotransferase) greater than (>)1.5 * upper limit of normal at screening
* Any loss of vision (permanent or transient blindness in 1 or both eyes, including ophthalmic migraine, transient ischemic attack, retinal artery/vein thrombosis)
* Known hereditary degenerative retinal disorders, including retinitis pigmentosa

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2021-08-08 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Analyte Concentration (Cmax) of Macitentan, its Metabolite ACT-132577, and Tadalafil | Predose and up to 216 hours post dose (Up to Day 10)
  Cmax is defined as maximum observed plasma analyte concentration.
Area Under the Concentration-time Curve from Time Zero to the Last Quantifiable Concentration (AUC [0-last]) of Macitentan, its Metabolite ACT-132577, and Tadalafil | Predose and up to 216 hours post dose (Up to Day 10)
  AUC(0-last) is the area under the plasma analyte concentration-time curve from time zero to time of the last quantifiable (non-below quantification limit [non-BQL]) concentration, calculated by linear-linear trapezoidal summation.
Area Under the Concentration-time Curve from Time Zero to Infinity (AUC [0-infinity]) of Macitentan, its Metabolite ACT-132577, and Tadalafil | Predose and up to 216 hours post dose (Up to Day 10)
  AUC (0-infinity) is the area under the analyte concentration-time curve (AUC) from time zero to infinite time, calculated as the sum of AUC (0-last) and C(last)/lambda(z); wherein AUC (0-last) is area under the plasma concentration-time curve from time zero to last measurable concentration, C(last) is the last observed measurable (non-BQL) analyte concentration; and lambda(z) is apparent terminal elimination rate constant.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Up to 8 weeks
  An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency